CLINICAL TRIAL: NCT05005611
Title: Probiotics Regulates Skin Care in Children : A Randomized, Double-blind Clinical Trial With Placebo
Brief Title: Probiotics Regulates Skin Care in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Glac Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Ho-Chang Kuo, Attending Physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: XPRPG8L0021~22; NCT05337670 (obsolete NCT alias)
Record Dates: First submitted 2021-08-10; First posted 2021-08-13 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Skin Care; Probiotics; Children

STUDY DESIGN:
Intervention Model Description: Skin Care in children.
Who Masked: Participant, Investigator
Masking Description: Double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Probiotics Lactobacillus salivarius AP-32 (Experimental)
  Interventions: Dietary Supplement: Probiotics Lactobacillus salivarius AP-32
- Probiotics Bifidobacterium animalis subsp. lactis CP-9 (Experimental)
  Interventions: Dietary Supplement: Probiotics Bifidobacterium animalis subsp. lactis CP-9
- Probiotics Lactobacillus rhamnosus LGG (Experimental)
  Interventions: Dietary Supplement: Probiotics Lactobacillus rhamnosus LGG

INTERVENTIONS:
Dietary Supplement: Placebo — A pack of powder without probiotics.
  1 pack / day
  Arms: Placebo
Dietary Supplement: Probiotics Lactobacillus salivarius AP-32 — A pack of powder with probiotics Lactobacillus salivarius AP-32
  1 pack / day
  Arms: Probiotics Lactobacillus salivarius AP-32
Dietary Supplement: Probiotics Bifidobacterium animalis subsp. lactis CP-9 — A pack of powder with probiotics Bifidobacterium animalis subsp. lactis CP-9
  1 pack / day
  Arms: Probiotics Bifidobacterium animalis subsp. lactis CP-9
Dietary Supplement: Probiotics Lactobacillus rhamnosus LGG — A pack of powder with probiotics Lactobacillus rhamnosus LGG
  1 pack / day
  Arms: Probiotics Lactobacillus rhamnosus LGG

SUMMARY:
Probiotics, a component that is generally referred to as a living microorganism or a microorganism present in a host. Most studies have shown that probiotics can regulate immune function in the body. Many studies have attempted to understand whether the use of probiotics can prevent allergic diseases or not.

ELIGIBILITY:
Inclusion Criteria:

* Estimated by PI.

Exclusion Criteria:

* Be allergic to medicine
* Take medicine like immune inhibition, or steroid injection in two weeks
* Participate in another clinical research or immune therapy in one month
* Have severe disease
* Inappropriate for this trial judged by PI

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin severity scoring | 3 months
  According to the scale to estimate skin severity

SECONDARY OUTCOMES:
Blood analysis | 3 months
  ELISA analysis
NGS in gastrointestinal tract | 3 months
  The difference of NGS ( Next Generation Sequence ) in gastrointestinal tract between 0 month and the 3rd month.
Life quality | 3 months
  The questionnaire of life quality in three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan